CLINICAL TRIAL: NCT01462279
Title: The Effect of Thiamine on VO2 Levels in Critically Ill Patients
Brief Title: Effect of Thiamine on Oxygen Utilization (VO2) in Critical Illness
Acronym: VO2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: American Medical Association (Other)
Responsible Party: Principal Investigator, Michael Donnino, Associate Professor of Emergency Medicine, Beth Israel Deaconess Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2010P000312
Record Dates: First submitted 2011-10-25; First posted 2011-10-31 (Estimated); Results first posted 2016-11-30 (Estimated); Last update posted 2018-01-16 (Actual); Status verified 2017-12

CONDITIONS: Acute Respiratory Failure
Keywords: acute respiratory failure; thiamine; oxygen consumption; VO2
MeSH Terms: interventions — Thiamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Thiamine (Experimental): Open label - 200mg IV
  Interventions: Drug: Thiamine

INTERVENTIONS:
Drug: Thiamine — 200mg of intravenous thiamine in 50ml of D5W will be infused over 30 minutes once

SUMMARY:
The objective of this study is to determine the effect of thiamine therapy on oxygen consumption in critically-ill patients. The investigators will evaluate this by measuring VO2 before and after thiamine administration in patients admitted to the ICU and requiring mechanical ventilation.

DETAILED DESCRIPTION:
Extensive research has been done over the past two decades looking at the role of oxygen delivery (DO2) and oxygen utilization (VO2) in critical illness. VO2 depends on cardiac output, arterial oxygen content, and the body's ability to extract oxygen effectively from the blood. Oxygen demand rises in critical illness as the body goes into a catabolic state, and lower VO2 has been associated with higher lactate levels and with poorer outcomes. Although increasing DO2 will often raise VO2, Hayes et al found that a subset of critically-ill patients failed to demonstrate a rise in VO2 in spite of achieving supranormal values of cardiac index (CI) and DO2. This group, in contrast to patients whose VO2 rose with the increase in CI and DO2, had exceedingly poor outcomes, suggesting that an inability to extract oxygen from the blood confers a poorer prognosis.(1)

Thiamine deficiency can manifest in several ways, but the syndrome of wet beriberi, caused by thiamine deficiency, includes lactic acidosis, cardiac decompensation and vasodilatory shock, similar to sepsis and other forms of critical illness. The mechanism by which thiamine deficiency causes dysfunction rests upon the vitamin's essential role in the Krebs cycle and Pentose Phosphate Pathway. Lack of adequate thiamine results in the failure of pyruvate to enter the Krebs Cycle, thus preventing aerobic metabolism. The resulting decrease in aerobic metabolism and increase in anaerobic metabolism leads to decreased oxygen consumption by the tissues and increased lactic acid production. The investigators group has found previously that upwards of 20% of critically ill patients with sepsis are thiamine deficient within 72 hours of presentation. In a dog model of septic shock, Lindenbaum et al have shown that, regardless of thiamine levels, supplementation with thiamine improved not only lactate clearance and mean arterial pressure, but increased VO2 as well. The effect of thiamine on VO2 in critically ill humans has not yet been reported, but an increase in VO2 max after administration of thiamine to healthy volunteers has been described. VO2 is known to rise in inflammatory states, reflecting increased energy expenditure. Prior studies have shown that VO2 will decrease with interventions such as fever control. In spite of VO2 being higher than normal in critically-ill patients, however, the end-organ damage and lactic acidosis suggest that it is not high enough to meet the metabolic demands of the critically-ill body. If the investigators were able to increase VO2 further in critically-ill patients, the investigators could potentially help maintain aerobic metabolism and decrease tissue hypoxia and the resulting end-organ damage. The investigators hypothesis is that administering thiamine intravenously to critically-ill patients will increase VO2.

Multiple methods of measuring VO2 have been used in the ICU, but in the current era where invasive monitoring with routine use of PA catheters is no longer the norm, indirect calorimetry became, for a time, the gold standard for measurement of gas exchange in critically ill, mechanically ventilated patients.(2) The metabolic cart used for indirect calorimetry is cumbersome and requires frequent calibration to maintain accuracy, however, and a newer, more portable method has been designed. The Datex-Ohmeda M-COVX device has been approved for the measurement of VO2 and VCO2 in mechanically ventilated patients. In studies, it has been validated as a method that is as accurate as indirect calorimetry, and perhaps even more accurate at higher FiO2.(3,4) The Datex-Ohmeda M-COVX connects to the Carescape B650 monitor made by GE, and measures VO2 through a single-use spirometer that attaches to the patient's ventilator tubing. In the following proposal, the investigators present a plan to examine the effect of thiamine therapy on VO2 in 30 critically-ill, mechanically ventilated patients, using the Datex-Ohmeda M-COVX module to measure VO2 before and after thiamine administration.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (age > 18 years) admitted to an ICU
* Mechanically ventilated

Exclusion Criteria:

* Unstable ventilator settings during measurement of VO2
* Temp > 100 at time of VO2 measurement
* FIO2 > 60%
* Endotracheal cuff leak, chest tube, or other evident source of air leak
* Thiamine supplementation within 24 hours prior to study enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2011-09; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Katherine M Berg, MD, Principal Investigator — Beth Israel Deaconess Medical Center; Michael W Donnino, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center (BIDMC), Boston, Massachusetts, United States

REFERENCES:
- [Derived] Berg KM, Gautam S, Salciccioli JD, Giberson T, Saindon B, Donnino MW. Intravenous thiamine is associated with increased oxygen consumption in critically ill patients with preserved cardiac index. Ann Am Thorac Soc. 2014 Dec;11(10):1597-601. doi: 10.1513/AnnalsATS.201406-259BC. PMID 25390455

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Thiamine
Started | 20
Completed | 17
Not Completed | 3

BASELINE CHARACTERISTICS:
Arm/Group | Thiamine
Number analyzed (Participants) | 17
Age, Continuous [Mean (Standard Deviation); unit: years] | 66 (17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 16
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 15
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 17

OUTCOME MEASURES:

1. Primary Outcome: Improvement in VO2
Description: VO2 measurements are taken at baseline and VO2 is continuously monitored over 9 hours. Thiamine is administered three hours after baseline measurements are taken.
Time Frame: Baseline to 9 Hours
Measure: Mean (Standard Deviation); unit: ml/min
Arm/Group | Thiamine
Number analyzed (Participants) | 17
ml/min | 16.9 (8.6)

2. Secondary Outcome: Improvement in Hemodynamics
Description: Hemodynamics were collected in all patients but we did not evaluate change in hemodynamics over the 9 hour protocol of the study. Due to the single-arm nature and small size of the study, and with no comparison arm, we did not think we had the statistical power to evaluate for a change in hemodynamics so this was not a planned outcome and was entered in error.
Time Frame: Baseline to Nine Hours
Population: Due to the single-arm nature and small size of the study, and with no comparison arm, we did not think we had the statistical power to evaluate for a change in hemodynamics so this was not a planned outcome and was entered in error.
Arm/Group | Thiamine
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Thiamine
Serious Adverse Events (participants affected / at risk) | 0/17
Other Adverse Events (participants affected / at risk) | 0/17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No